CLINICAL TRIAL: NCT04568876
Title: Efficacy of Palmitoylethanolamide, in add-on to Standard Therapy, on Inflammatory Markers of Patients With Interstitial Pneumonia Due to COVID-19. A Pilot Controlled, Randomized, Open Lable Clinical Study
Brief Title: Micronized and Ultramicronized Palmitoylethanolamide in COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epitech Group SpA (Industry)
Collaborators: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NORM_MPS-COVID; NORM_MPS_11 (Other: Epitech Group)
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Suspensions; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEA Group (Active Comparator): Normast® MPS (mPEA and umPEA 300mg + 600mg) oral suspension: 2700mg/die in 3 doses for 28 days, in add-on to standard therapy
  Interventions: Dietary Supplement: Micronized and ultra-micronized Palmitoylethanolamide (mPEA and umPEA, 300mg + 600mg) oral suspension; Combination Product: Standard Therapy
- Control Group (Other): Standard therapy only
  Interventions: Combination Product: Standard Therapy

INTERVENTIONS:
Dietary Supplement: Micronized and ultra-micronized Palmitoylethanolamide (mPEA and umPEA, 300mg + 600mg) oral suspension — Micronized and ultra-micronized Palmitoylethanolamide is on the market in Italy as a Food for Special Medical Purposes
  Other Names: Normast® MPS oral suspension
  Arms: PEA Group
Combination Product: Standard Therapy — Standard therapy established for individual patients

SUMMARY:
SARS-CoV-2 infection is a condition characterized by excessive leukocyte infiltration, massive release of chemokines, proteases and cytokines, the so-called "cytokine storm", which promote the inflammatory process and contribute to exacerbation of COVID-19 symptomatology. Because of the abnormal release of pro-inflammatory cytokines by non-neuronal cells of the immune system, such as the mast cells in periphery, and microglia at central level, the body activates a defensive neuroinflammatory process that, if not controlled, can become pathological. Therefore it's important to intervene early on neuroinflammation, in order to limit the progression of the disease.

A possible intervention is represented by Palmitoylethanolamide (PEA), an endogenous molecule of the N-acylethanolamine family synthesized "on demand" in response to "stress factors" to restore tissue homeostasis, able to control mast cells and microglia uncontrolled activation. Experimental evidence in vitro and in vivo demonstrated the anti-inflammatory and neuroprotective effect of micronized and ultra-micronized PEA (mPEA and umPEA), confirmed in various clinical investigations conducted in patients with different pathological conditions. The aim of this study is to investigate the efficacy of a compound containing mPEA + umPEA on peripheral inflammatory markers, neuroinflammation, and others clinical parameters in intensive care patients with COVID-19 interstitial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Unit Hospitalization for interstitial pneumonia due to COVID-19 diagnosis (nasal swab/sputum/bronchoalveolar lavage positive for Sars-Cov-2 infection)

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Known allergy or hypersensitivity to the product or its excipients;
* Inability to take the product per os or via nasogastric tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Number of responder participants after 7 days of treatment | 7 days
  Responder: decrease ≥ 30% from baseline of IL-6 blood levels

SECONDARY OUTCOMES:
Change of pro-inflammatory markers (IL-6, IL-1 alpha, IL-1 beta, TNF-alpha, PCR, PCT, neopterin) | 0, 3, 7, 14, 28 days
Change of anti-inflammatory markers (IL-4, IL-10) | 0, 3, 7, 14, 28 days
Change of brain damage markers (S100b, ENS) | 0, 3, 7, 14, 28 days
Change of coagulation indices (INR, fibrinogen, D-dimer) | 0, 3, 7, 14, 28 days
Change of hematological parameters | 0, 3, 7, 14, 28 days
  leukocyte formula (lymphocytes, CD4 / CD8 ratio)
Change of oxygenation indices (P/F ratio, lactates) | 0, 3, 7, 14, 28 days
Number of participants who developed delirium | 0, 3, 7, 14, 28 days
  Confusion Assessment Method-Intensive Care Unit (CAM-ICU) (0-1: no delirium; >1 delirium)
Number of participants who developed anxiety and/or depression | 0, 3, 7, 14, 28 days
  Hospital Anxiety and Depression Scale (HADS) (0: normal; 21: severe)

OTHER OUTCOMES:
Number of days of invasive mechanical ventilation (orotracheal intubation - IOT) | 28 days
Number of days of non-invasive mechanical ventilation (Helmet, face mask) | 28 days
Number of days of intensive care (ICU) hospitalization | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof.ssa Flaminia Coluzzi, MD, Principal Investigator — Azienda Ospedaliera Universitaria Sant'Andrea di Roma
Locations (1):
- Anestesia e Rianimazione Azienda Ospedaliera Universitaria Sant'Andrea, Roma, Italy